CLINICAL TRIAL: NCT00227058
Title: Effects of Orotic Acid Derivatives With or Without Glutathione on Allergic
Brief Title: Effects of Orotic Acid Derivatives With or Without Glutathione on Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Kyowa Hakko Kogyo Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KHK040213
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Orotic Acid

INTERVENTIONS:
Drug: Orotic acid and Glutathione-(Nutritional Supplements)

SUMMARY:
The purpose of this study is to learn if two nutritional supplements, Orotic Acid and Glutathione will have any effect on the immune system response and if there will be any effect on the symptoms of seasonal allergies. It is our thinking that they will have an positive effect.

DETAILED DESCRIPTION:
Current therapy for most immune-based diseases center around the use of anti inflammatory agents, many of which have unpleasant or dangerous side effects. Allergic rhinitis affects over 40 million Americans and its morbidity results from a combination of physical and psychological symptoms. The primary immunopathology has been defined as an imbalance of TH1/TH2 cytokines production resulting in increased allergen-specific IgE production, mast cell activation and eosinophil recruitment/activity. Metallic salts of orotic acid (OR), a natural intermediate in pyrimidine nucleic acid synthesis have been utilized to improve the signs and symptoms of a variety of maladies including the common cold, allergies and as preventatives for cancer and heart disease. Recent studies have reported that moderate doses of OR can mitigate or prevent endocrine and subjective psychological stresses in an acute laboratory stress model. All these findings lead us to hypothesize that OR salts administration will alleviate or eliminate the signs and symptoms associated with seasonal AR through a protective effect that involves direct anti-inflammatory immune effects and/or immunomodulation that include leukocyte trafficking, immunoregulatory cytokine balance and/or decrease inflammatory cell activity.

ELIGIBILITY:
Inclusion Criteria: Participants must have allergic rhinitis and be skin test positive to Bermuda Grass, Johnson grass, oak tree and/or ragweed, be symptomatic -

Exclusion Criteria: Any significant known heath disease: cardiovascular disease, cancer, or any metabolic disorder, smoker

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2005-01; Study Completion 2005-11

PRIMARY OUTCOMES:
Improvement in nasal symptom scores from baseline after intervention

SECONDARY OUTCOMES:
change in cytokine profile with intervention compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D. Marshall, MD/PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States